CLINICAL TRIAL: NCT04060459
Title: Paclitaxel-binding Albumin and Cisplatin as Neoadjuvant Chemotherapy in Patients With Muscle-Invasive Bladder Cancer - A Single-center, Single-arm and Stage II Clinical Study
Brief Title: Paclitaxel-binding Albumin and Cisplatin as Neoadjuvant Chemotherapy in Patients With Muscle-Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dong Wang, chief physician, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThirdMMUa
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2018-10

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer；Paclitaxel-binding albumin；Cisplatin；Neoadjuvant Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment plan (Experimental): Paclitaxel-binding albumin 260 mg/m2，d1，ivgtt；cisplatin 75 mg/m2，d1，ivgtt
  Interventions: Drug: Paclitaxel-binding albumin

INTERVENTIONS:
Drug: Paclitaxel-binding albumin — Paclitaxel-binding albumin 260 mg/m2，d1，ivgtt；cisplatin 75 mg/m2，d1，ivgtt

SUMMARY:
This is a phase II study of Paclitaxel-binding albumin, Cisplatin as neoadjuvant chemotherapy in patients with muscle-invasive urothelial carcinoma of the bladder. Patients with muscle invasive urothelial carcinoma who are candidates for radical cystectomy will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients must have histologically confirmed resectable（stage T2，T3 and T4a） urothelial carcinoma following 2017 V8 AJCC，including renal pelvic carcinoma，ureteral carcinoma，bladder carcinoma and urethral carcinoma.
3. There was at least one measurable tumor lesion following RECIST 1.1.
4. Treatment naïve.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. Left ventricular ejection fraction≥50%.
7. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L，platelets (PLT) ≥ 100 × 109/L，hemoglobin (Hb) ≥ 90 g/L，leucocyte ≥ 3.0 × 109/L.
8. Total bilirubin (TBIL) ≤ 1.5 ×institutional upper limit of normal (ULN)， Alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) /Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]≤ 2.5 ×ULN ，Creatinine (CRE) ≤ 1.5 ×ULN.
9. Signed informed content obtained prior to treatment.

Exclusion Criteria:

1. Patients who are pregnant or may be pregnant or nursing.
2. Patients with Coagulation dysfunction or active internal hemorrhage.
3. Patients with uncontrolled active infection，HIV，viral hepatitis.
4. Peripheral nerve lesion≥grade 1 following NCI-CTC 5.0.
5. Patients with serious cardiovasculardisease including history of cerebral vascular accident ， myocardial infarction，hypertension，angina，heart failure（NYHA grade 2-4） within the last 6 months.
6. History of allergic reactions attributed to compounds of similar chemical or biological composition to drugs used in this study.
7. Patients was involved in another study within the last 30 days.
8. Patients was mental disorders.
9. Any other patients deemed by the attending physician to be unsuitable to allow the feasible for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The Pathologic Complete Response Rate (<pT0) of Neoadjuvant Paclitaxel-binding albumin and Cisplatin in Patients With Muscle-invasive Bladder Cancer. | 2 years
  Complete pathologic response to neoadjuvant GCS is the primary endpoint is defined as the absence of carcinoma (pT0 disease) and the absence of microscopic lymph node metastases (N0) on the final cystectomy specimen.

SECONDARY OUTCOMES:
The Pathologic Response Rate (<pT2) of Neoadjuvant Paclitaxel-binding albumin and Cisplatin in Patients With Muscle-invasive Bladder Cancer. | 2 years
  is defined as the absence of muscle invasive carcinoma (<pT2 disease) and the absence of microscopic lymph node metastases (N0) on the final cystectomy specimen

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, Principal Investigator — Daping Hospital, Third Military Medical University, Chongqing,China
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided